CLINICAL TRIAL: NCT04281953
Title: Long-term Ototoxicity in Cancer Survivors Treated With Chemotherapy and the Impact on Quality of Life
Brief Title: Impact on Quality of Life of Long-term Ototoxicity in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); International Stem Cell Forum (Other)
Responsible Party: Sponsor
Other Study IDs: 18074
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Quality of Life; Cancer; Hearing Loss, Sensorineural; Tinnitus, Subjective; Late Effect
MeSH Terms: conditions — Neoplasms; Hearing Loss, Sensorineural; Tinnitus | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with ototoxicity: People living with and beyond who experience ototoxicity as a result of chemotherapy
  Interventions: Diagnostic Test: High frequency audiometry; Other: Short-Form 36-Item Questionnaire (SF-36); Other: Hearing handicap inventory for adults/elderly (HHIA/HHIE); Other: Tinnitus handicap inventory (THI)

INTERVENTIONS:
Diagnostic Test: High frequency audiometry — Simple hearing test
Other: Short-Form 36-Item Questionnaire (SF-36) — Questionnaire on quality of life (Short Form 36 Item- SF-36)
Other: Hearing handicap inventory for adults/elderly (HHIA/HHIE) — Questionnaire on Hearing loss (Hearing handicap inventory for adults/elderly- HHIA/HHIE)
Other: Tinnitus handicap inventory (THI) — Questionnaire on Tinnitus (Tinnitus Handicap Inventory)

SUMMARY:
This project aims to explore, in depth, the burden of hearing loss and tinnitus on cancer survivors. Using semi-structured interviews, audiograms and a variety of validated questionnaires, the specific impact ototoxicity has on quality of life will be investigated.

From this, we can identify the specific needs of patients experiencing hearing loss and tinnitus following chemotherapy and develop a tailored and personalised support system.

DETAILED DESCRIPTION:
The medical and technological advances in cancer research have caused a decline in cancer deaths in recent decades. For example, the 5-year survival rate now is above 80% for many adult cancers, including breast and testicular cancers. In breast cancer alone, the mortality rate has reduced 39% since 1989 and currently has a 5 year survival rate over 90%. Due to this increase in survival rates and the intensity of treatment, many face long-term physical and psychological challenges in survivorship. Cancer survivors may experience altered body image and changes in sexual health and energy levels in addition to distress, anxiety, the fear of recurrence and the chronic side effects of their treatment. The need to research the long-term effects of chemotherapy and the impact they have on quality of life is crucial.

There is a need to broaden research beyond the survival rates and address the need for support for those who are adapting to a life after cancer. Survivors are left with often permanent and possible life-debilitating effects from treatment. To date, there has been little research on the specific late effects of chemotherapy and the associated impact on quality of life.

Platinum-based chemotherapy, although highly effective, is known to cause ototoxicity, presenting often as permanent high frequency hearing loss and tinnitus. Hearing loss and tinnitus are associated with a higher risk of depression, social isolation and anxiety. The quality of social interactions for a person with hearing loss and tinnitus is diminished as taking part in conversations becomes challenging. This is particularly problematic as it means that the quality of life of these cancer survivors is reduced.

The impact hearing loss and tinnitus has on quality of life in cancer survivors remains unclear and under-studied. Because cancer therapies can potentially cause life-threatening side effects such as cardiotoxicity and nephrotoxicity, these become the priority. However, once these side acute effects subside, other long-term side effects remain and can permanently reduce quality of life. Cancer survivors may have already experienced a difficult journey from the diagnosis itself, the physical challenges of treatment and finally, remission. Re-adapting back to their previous life whilst in remission, but with added permanent side effects, both physically and psychologically, can be extremely difficult for some survivors.

Currently, there is little information and support offered to these patients who suffer from ototoxicity, potentially leading to many being undiagnosed and untreated. These patients can be affected by this toxicity for the rest of their lives, which can have a detrimental impact on their quality of life. It is essential that a deeper understanding and increased awareness of how hearing loss and tinnitus affects the quality of life of cancer survivors is sought to improve long-term symptoms management and support offered. This study aims to develop this and improve the support given to cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Has had platinum-based chemotherapy between 0-5 years ago
* Has had at least 1 cycle- Was an adult (over 18) at the time of cancer diagnosis

Exclusion Criteria:

* Pre-existing hearing issues
* Radiotherapy to the head and neck area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have received platinum-based chemotherapy 0-5 years ago.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of hearing loss | Between 0-5 years
  High frequency audiogram

SECONDARY OUTCOMES:
Quality of life Questionnaire SF-36 (short-form 36 item) | Between 0-5 years
  Questionnaire on quality of life, scale between 0-100 with 0 being bad quality of life and 100 being good
Hearing Questionnaire HHIA/HHIE (hearing handicap inventory for adults/elderly) | Between 0-5 years
  Questionnaire on hearing loss scale from 0-100, 0 being no handicap and 100 being a big handicap
Tinnitus Questionnaire THI (tinnitus handicap inventory) | Between 0-5 years
  Questionnaire on Tinnitus from 0-100, 0 being no handicap and 100 being a bit handicap

CONTACTS AND LOCATIONS:
Overall Officials: David Baguley, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be anonymised and made confidential, statistical analysis will be performed before data is shared.